CLINICAL TRIAL: NCT03595839
Title: Fistuolotomy With or Without Marsupialization for Treatment of Simple Anal Fistula: a Randomized Controlled Trial
Brief Title: Fistulotomy With or Without Marsupialization for Treatment of Simple Anal Fistula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Lecturer of general surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: mansoura60
Record Dates: First submitted 2018-07-11; First posted 2018-07-23 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Anal Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fistulotomy with Marsupialization (Active Comparator): Lay open and Marsupialization of the fistula track
  Interventions: Procedure: Fistulotomy; Procedure: Marsupialization
- Fistulotomy without Marsupialization (Active Comparator): lay open of the fistula track
  Interventions: Procedure: Fistulotomy

INTERVENTIONS:
Procedure: Fistulotomy — The fistula track is laid open after complete probing till the internal opening
Procedure: Marsupialization — The laid open track will be marsupialized using interrupted absorbable sutures
  Arms: Fistulotomy with Marsupialization

SUMMARY:
Patients with simple anal fistula will undergo fistulotomy operation and will be divided into two groups: the first will undergo marsupialization of the laid open fistula track and second group will not undergo marsupialization. The effect of marsupialization on healing of anal fistula will be compared postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Age: 18-65 years
* All Patients with primary simple anal fistula (subcutaneous, intersphincteric, or low trans-sphicnteric involving less than 25% of external anal sphincter fibers).

Exclusion Criteria:

* High trans-sphincteric, extra-sphincteric, supra-sphincteric, secondary.
* Recurrent anal fistulas.
* Patients associated with anorectal pathology such as anal fissure, hemorrhoids, rectal prolapse, neoplasm, solitary rectal ulcer, inflammatory bowel diseases and TB.
* High risk patients according to ASA (American society of anesthesiologists )
* Any degree of incontinence.
* Patients with previous anal surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Time to complete healing | 8 weeks
  The duration of time required to achieve complete wound healing

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Emile, M.D., Principal Investigator — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No